CLINICAL TRIAL: NCT05405634
Title: Microbiota in Chronic Anal Fissure and Its Association With Prognosis - Prospective Cohort Study
Brief Title: Microbiota in Chronic Anal Fissure and Its Association With Prognosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Lasse Krogsbøll (Other)
Responsible Party: Sponsor-Investigator, Lasse Krogsbøll, Sponsor-investigator, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Other Study IDs: Microbiota in anal fissure
Record Dates: First submitted 2022-05-20; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Anal Fissure; Microbial Colonization
MeSH Terms: conditions — Fissure in Ano; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Swab from anal fissure/anoderm and rectum, and tissue removed by fissurectomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with chronic analfissure: 1. Consecutive patients referred to the outpatient clinic at the Digestive Disease Centre, Bispebjerg Hospital in Denmark for botox injection for chronic anal fissure. Thus, the included patients will likely all have tried conservative treatment before referral, and are expected to represent a more homogeneous subset with longer standing disease, less spontaneous improvement, and a higher likelihood of being compliant with suggested therapy
- Patients with an indication for fissurectomy: Consecutive patients with an indication for revision of the fissure and anal injection of botulinum toxin in general anaesthesia
- Healthy volunteers: Healthy volunteers. These will be recruited among staff at the Digestive Disease Centre, Bispebjerg Hospital, Denmark.

SUMMARY:
In this study, we will try to answer the following questions:

1. What are the salient features of the microbiota in chronic anal fissure?
2. Are these features associated with prognosis and response to therapy?
3. Does an anal fissure swab and anal fissure tissue give comparable bacteriological results?

DETAILED DESCRIPTION:
To allow rational planning of therapeutic trials of antimicrobial or biofilm degrading medical therapy, a better understanding of the microbiota of chronic anal fissures is needed. Previous studies have relied on culture, whereas we will employ molecular methods.

We will collect bacteriological samples from patients referred to us with anal fissure, in order to characterize the microbiota. To see if the microbiota is distinct from or similar to the rectal microbiota, we will also collect a swap from the rectum. We will also collect swaps from the anal verge of healthy volunteers without anal fissure, to see if the microbiota in anal fissures are distinct from the normal anodermal microbiota. To examine whether a swap is a reliable method for characterizing the microbiota in anal fissure, we will also collect excised anal fissure tissue from the subset of patients with a clinical indication for fissurectomy in general anaesthesia, and compare the analysis results with those from the swap.

We will re-assess the patients clinically and with a repeat swap after 3 months, and perform an exploratory analysis in order to identify possible features of the microbiota that are associated with poor response to therapy.

ELIGIBILITY:
Inclusion criteria

Three samples will be included:

1. Consecutive patients referred to the outpatient clinic at the Digestive Disease Centre, Bispebjerg Hospital in Denmark for botox injection for chronic anal fissure. Thus, the included patients will likely all have tried conservative treatment before referral, and are expected to represent a more homogeneous subset with longer standing disease, less spontaneous improvement, and a higher likelihood of being compliant with suggested therapy
2. Consecutive patients with an indication for revision of the fissure and anal injection of botulinum toxin in general anaesthesia
3. Healthy volunteers. These will be recruited among staff at the Digestive Disease Centre, Bispebjerg Hospital, Denmark.

Samples 1 and 2 will not be independent, as patients from group 1 may be included in group 2 depending on the clinical course. No direct comparisons between these two groups are planned (see analysis section).

Exclusion criteria

* Symptom duration of less than 8 weeks (groups 1 and 2)
* Known or suspected Crohn's disease
* Known or suspected active venereal disease.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: As above.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
16S/18S RNA | Baseline
16S/18S RNA | 3 months
PICRUSt2 | Baseline
PICRUSt2 | 3 months
Healing of anal fissure after 3 months | 3 months
  Defined by complete patient-reported resolution of pain combined with healed fissure on clinical examination
Change from baseline in pain severity both during and after defecation | 3 months
  Numerical rating scale 1-10.

CONTACTS AND LOCATIONS:
Overall Officials: Lasse T Krogsbøll, MD, PhD, Principal Investigator — Digestive disease center, Bispebjerg Hospital

IPD SHARING:
Plan to Share IPD: Undecided